CLINICAL TRIAL: NCT05749276
Title: Multicentric Phase 1 Study With Escalation of Doses of Daratumumab in Combination With Chemotherapy (Idarubicin and Cytarabine) in Patients of 60 Years Old or More With Adverse Risk Acute Myeloblastic Leukemia (AML) (DARALAM)
Brief Title: Escalation of Doses of Daratumumab in Combination With Chemotherapy (Idarubicin and Cytarabine) in Patients of 60 Years Old or More With Adverse Risk Acute Myeloblastic Leukemia (AML) (DARALAM)
Acronym: DARALAM
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC22_0372
Record Dates: First submitted 2023-02-13; First posted 2023-03-01 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Adult Patients With Adverse Risk Acute Myeloblastic Leukemia
MeSH Terms: interventions — daratumumab

STUDY DESIGN:
Intervention Model Description: Continual Reassessment Method for MTD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Darzalex (Experimental): DARZALEX®
  Dose level 1 : 1800 mg Day 1 Dose level 2 : 1800 mg Day 1 and 8 (+/- 2 days) Dose level 3 : 1800 mg à Day 1, 8 (+/- 2 days) and D15 (+/- 2 days)
  Interventions: Drug: Darzalex

INTERVENTIONS:
Drug: Darzalex — DARZALEX® = Daratumumab. Solution for injection, 1800 mg/15 mL, single vial. Sub-cutaneous administration.
  * Dose level 1 : 1800 mg Day 1
  * Dose level 2 : 1800 mg Day 1 and 8 (+/- 2 days)
  * Dose level 3 : 1800 mg à Day 1, 8 (+/- 2 days) and D15 (+/- 2 days)

SUMMARY:
To search for a Maximum Tolerated Dose (MTD) for the combination of daratumumab and induction chemotherapy with Idarubicin and cytarabine in patients with Acute Myeloblastic Leukemia (AML) of poor prognosis

ELIGIBILITY:
Inclusion Criteria:

* Age >= 60 ans
* Poor prognosis AML defined according to the following criteria:1. For first-line AML:intermediate or unfavorable risk according to ELN 2022 2.for Relapsed AML:regardless of the ELN risk group
* ECOG <= 2
* Patient eligible for intensive chemotherapy
* Who provide their written informed consent
* Liver workup: transaminases < 3x normal, bilirubin < 1.5 X normal
* Creatinine clearance > 60ml/mn
* LVEF >= 50%.

Exclusion Criteria:

* Patients with FLT3 ITD or TKD mutation
* Patients with tuberculosis
* Patients with documented active infection with COVID 19
* Patients with hereditary fructose intolerance (HFI)
* Uncontrolled infection
* Active or past infection with Hep B, C or HIV+
* Not Affiliated with French social security system or no beneficiary from such system
* Pregnant women or patients who cannot take contraception ( contraceptive pill, abstinence, unauthorised IUD) in case of fertility. A patient who cannot continue contraception for at least 6 months after the last injection of DARATUMUMAB is not eligible for inclusion.
* Breastfeeding women
* Minors
* Adults under guardianship, curatorship or safeguard of justice
* Hypersensitivity to any of the active ingredients or excipients
* Patients with significant cardiovascular pathology including any of the following: myocardial infarction within 6 months prior to study entry, unstabilized coronary artery disease, uncontrolled hypertension, congestive heart failure.
* Patient with disease requiring systemic immunosuppressive therapy (such as high-dose steroids defined as ≥ 10mg prednisone or equivalent per day) within 4 weeks prior to the 1st scheduled dose of study treatment with the exception of dermocorticoids

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
DLT | DAY 45
  Dose at which no toxic effect is observed, by determination of the LDT (Toxic Limit Dose). A TLD is defined by the occurrence of grade ≥ 3 daratumumab related toxicity that is not reversible after 7 days (except for haematological toxicity) or the absence of emergence from aplasia at D45 of induction (in the absence of treatment failure). Toxicity is assessed according to NCI-CTCAE version 5 criteria. The search for DLT is continued until D45 of induction.

SECONDARY OUTCOMES:
response to the induction treatment | DAY 45
  calculation of the rate of complete remission (CR) with negative residual disease (CR MRD-), CR, CR with incomplete haematological recovery (CRi), MLFS (morphological leukemia free state), partial response (PR) or treatment failure according to the 2022 NLE definition between D30 and D45.
Assessment of myelotoxicity | Day 1
  Neutrophil recovery time (>1.0 × 109/L) from D1 - Recovery time of platelets (>100 × 109/L) from D1
Overall survival (OS) | 6 months
  time from D1 of induction to date of last contact or death
Event-free survival (EFS) | 6 months
  time from D1 of induction to date of relapse, death or date of last
Relapse incidence | 6 months
Flow cytometry (FCM) investigation of myeloid-derived suppressor cells | Day 45
Comparison of MDSC values in CMF | Day 45
research on the level of CD38 expression on blasts | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: MATHILDE HUNAULT, Principal Investigator — University Hospital, Angers; MARC BERNARD, Principal Investigator — CHU Rennes